CLINICAL TRIAL: NCT06980701
Title: Improving Oral and Systemic Health in Individuals With Prediabetes Through Personalized Oral Hygiene Advice Provided by Dentists or by Artificial Intelligence: A Randomized Clinical Trial
Brief Title: Improving Oral and Systemic Health in Individuals With Prediabetes Through Personalized Oral Hygiene Advice Provided by Dentists or by AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Walter Y.H. Lam, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 24-658
Record Dates: First submitted 2025-05-01; First posted 2025-05-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Gum Disease; Prediabetes
Keywords: gum disease; prediabetes; oral health; oral hygiene
MeSH Terms: conditions — Gingival Diseases; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI OHI group (Experimental): Personalized oral hygiene instructions provided by AI on the adequacy of patients' home care.
  Interventions: Behavioral: AI OHI group
- Dental professionals OHI group (Active Comparator): Personalized oral hygiene instructions provided by a dental professional on the adequacy of patients' home care
  Interventions: Behavioral: Dental professionals OHI group

INTERVENTIONS:
Behavioral: AI OHI group — The participants will receive personalized OHI such as toothbrush and interdental cleaning to specific areas provided by AI. An mHealth system will be used to detect intraoral photograph of anterior teeth and analysis of the photograph and label the gum condition as Healthy (green)/questionable (yellow)/diseased (red) within 2 minutes by AI. Then specific OHI to each particular site would be provided by AI according to tested results on the photograph
  Other Names: AI
  Arms: AI OHI group
Behavioral: Dental professionals OHI group — ll participants will receive personalized OHI by dental professionals. This instruction includes brushing and interdental cleaning in each particular dental site. If they have any personal concern or unclear points regarding oral hygiene practice, they can ask.
  Other Names: conventional OHI
  Arms: Dental professionals OHI group

SUMMARY:
Prediabetes is an intermediate stage before the development of diabetes, characterized by elevated blood glucose levels but lower than the diagnostic criteria of diabetes and is associated with multiple long-term complications. This systemic disease is mutually linked to inflammatory gum diseases through circulating inflammatory mediators. Controlling inflammatory gum diseases improves blood glucose levels and reduces long-term complications. While maintaining good oral hygiene through home care is essential for managing inflammatory gum diseases, close supervision of patients' home care is labor-intensive and expensive. Artificial Intelligence (AI) has been used to provide personalized advice on the adequacy of patients' home care (oral hygiene). The investigators hypothesize that the use of AI can improve home care, thereby enhancing both gum health and systemic health, similar to human dental professionals.

DETAILED DESCRIPTION:
Prediabetes is an intermediate stage before the development of diabetes, characterized by elevated blood glucose levels but lower than the diagnostic criteria of diabetes and is associated with multiple long-term complications. This systemic disease is mutually linked to inflammatory gum diseases through circulating inflammatory mediators. The relation between oral health and prediabetes management has long been under-appreciated. People with prediabetes have a 2-3-fold greater risk for periodontitis compared to people without prediabetes. The progression and severity of periodontitis are also greater in prediabetic patients. According to the National Health and Nutrition Examination Survey, the severity of periodontitis is positively associated with the risk as well as the prevalence of prediabetes. A growing body of data indicates that oral inflammation has an impact on general diseases. Controlling inflammatory gum diseases improves blood glucose levels and reduces long-term complications. While maintaining good oral hygiene through home care is essential for managing inflammatory gum diseases, close supervision of patients' home care is labor-intensive and expensive.

Nowadays, artificial intelligence (AI) can readily assist in the self-detection of diseases, including gum disease, allowing older adults to identify diseases early and prevent further complications. The use of AI-based mHealth has become increasingly effective in promoting periodontal health by adopting simple, AI-driven self-tests using smartphones. Another systematic review done by investigators' team found that AI-based mHealth for oral hygiene and gum disease monitoring showed clinical effectiveness across different clinical scenarios. The investigators' team has already launched an AI system for the detection of gum disease using smartphone intraoral photography, in which the system can detect colour changes of gum inflammation in specific sites in intraoral photography and diagnose as three simple situations (severe, mild and no inflammation). The AI system have high sensitivity 92% to identify disease from sites that have gingivitis, and high specificity 94% to identify healthy tissue from sites that have no gingivitis using professional intraoral photography. Moreover, the investigators have tested that the accuracy of colour captured by a smartphone is comparable to that captured by a professional single-lens reflective camera. The investigators' team already have applied the AI-powered smartphone photography among 38 older adults in 5 day-care centres of Hong Kong to test participants' gum health. The result is promising with accuracy of 96% sensitivity and 82% specificity. The present study will apply AI technology on disease detection and giving personalized oral health instruction (OHI) closely to the patients to maintain periodontal health and consequently prediabetic control.

In this study, the hypothesis is that the use of AI can improve home care, thereby enhancing both gum health and systemic health, similar to human dental professionals.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects who are >18 years of age and able to give informed consent.
* - Subjects who are mentally and cognitively healthy.
* - Subjects who have at least 6 anterior maxillary or mandibular natural teeth including incisors and canine.
* - Subjects who are with prediabetic state with impaired HbA1c 5.7% to 6.4%, impaired fasting plasma glucose level 5.6mmol/L to 6.9 mmol/L and/or impaired plasma glucose level after 2h OGTT 7.8 mmol/L to 11.0 mmol/L.
* - Subjects who can speak, read, or understand Cantonese to complete the satisfaction questionnaire.
* - Subjects who can practice oral hygiene procedure (regular tooth brushing and interdental cleansing/flossing/brushing) daily on their own independently.

Exclusion Criteria:

* - Subjects who have less than 6 anterior maxillary or mandibular natural teeth with or without dental prostheses in those area.
* - Subjects who are with a current diagnosis or clinical history of T2DM.
* - Subjects who have mental illness, or similar problems that unable to complete the satisfaction questionnaire.
* - Subjects who cannot perform oral hygiene procedure (regular tooth brushing and interdental cleansing/flossing/brushing) by any condition of oral cavity such as tumor or maxillomandibular fixation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Gum inflammation at baseline | baseline
  Gum inflammation will be evaluated using BPE score (from 0 to 4), which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group)
Gingival health at baseline | baseline
  Gingival health will be assessed by gingival index (Löe H 1967), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group)
Oral hygiene status at baseline | baseline
  Oral hygiene status will be assessed by plaque index (Silness and Loe, 1965), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group)
HbA1c level at baseline | baseline
  Glycaemic level at baseline is evaluated by HbA1c level (glycated haemoglobin that measures glycaemic control over the past 2-3 months). Prediabetes is defined as HbA1c of 5.7-6.4% (39-47 mmol/mol)
FPG level at baseline | baseline
  Glycaemic level at baseline is evaluated by FPG (fasting plasma glucose level that measures the blood sugar levels). Prediabetes is defined as 100-125 mg/dL (5.6-6.9 mmol/L)
2-h PG during 75-g OGTT level at baseline | baseline
  Glycaemic level at baseline is evaluated by 2-h PG during 75-g OGTT (plasma glucose level after 2-hour 75-g oral glucose tolerance test). Prediabetes is defined as 2-h PG during 75-g OGTT of 140-199 mg/dL (7.8-11.0 mmol/L)
Gum inflammation at 3-month | 3-month
  Gum inflammation will be evaluated using BPE score (from 0 to 4), which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 3-month follow up
Gingival health at 3-month | 3-month
  Gingival health will be assessed by gingival index (Löe H 1967), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 3-month follow-up
Oral hygiene status at 3-month | 3-month
  Oral hygiene status will be assessed by plaque index (Silness and Loe, 1965), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 3-month follow-up
HbA1c level at 3-month | 3-month
  Glycaemic level at 3-month follow-up is evaluated by HbA1c level (glycated haemoglobin that measures glycaemic control over the past 2-3 months). Prediabetes is defined as HbA1c of 5.7-6.4% (39-47 mmol/mol)
FPG level at 3-month | 3-month
  Glycaemic level at 3-month follow-up is evaluated by FPG (fasting plasma glucose level that measures the blood sugar levels). Prediabetes is defined as 100-125 mg/dL (5.6-6.9 mmol/L)
2-h PG during 75-g OGTT level at 3-month | 3-month
  Glycaemic level at 3-month follow-up is evaluated by 2-h PG during 75-g OGTT (plasma glucose level after 2-hour 75-g oral glucose tolerance test). Prediabetes is defined as 2-h PG during 75-g OGTT of 140-199 mg/dL (7.8-11.0 mmol/L)
Gum inflammation at 9-month | 9-month
  Gum inflammation will be evaluated using BPE score (from 0 to 4), which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 9-month follow up
Gingival health at 9-month | 9-month
  Gingival health will be assessed by gingival index (Löe H 1967), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 9-month follow-up
Oral hygiene status at 9-month | 9-month
  Oral hygiene status will be assessed by plaque index (Silness and Loe, 1965), with a scale from 0 to 3, which will be examined by a blinded assessor (a calibrated dentist who blinded to participants' group) at 9-month follow-up
HbA1c level at 9-month | 9-month
  Glycaemic level at 9-month follow-up is evaluated by HbA1c level (glycated haemoglobin that measures glycaemic control over the past 2-3 months). Prediabetes is defined as HbA1c of 5.7-6.4% (39-47 mmol/mol)
FPG level at 9-month | 9-month
  Glycaemic level at 9-month follow-up is evaluated by FPG (fasting plasma glucose level that measures the blood sugar levels). Prediabetes is defined as 100-125 mg/dL (5.6-6.9 mmol/L)
2-h PG during 75-g OGTT level at 9-month | 9-month
  Glycaemic level at 9-month follow-up is evaluated by 2-h PG during 75-g OGTT (plasma glucose level after 2-hour 75-g oral glucose tolerance test). Prediabetes is defined as 2-h PG during 75-g OGTT of 140-199 mg/dL (7.8-11.0 mmol/L)

SECONDARY OUTCOMES:
C-reactive protein level at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Inflammatory markers, i.e., C-reactive protein from serum, saliva and plaque samples (pg/mL) will be assessed at baseline, 3-month and 9-month follow-ups
IL6 level at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Inflammatory markers, i.e., IL6 from serum, saliva and plaque samples (pg/mL) will be assessed at baseline, 3-month and 9-month follow-ups
IL8 level at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Inflammatory markers, i.e., IL8 from serum, saliva and plaque samples (pg/mL) will be assessed at baseline, 3-month and 9-month follow-ups
Body weight at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Body weight (measured with standard procedures, in kilograms) will be assessed at baseline, 3-month and 9-month follow-ups
Percentage body fat at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Percentage body fat (using bioelectrical impedance analysis, %) will be assessed at baseline, 3-month and 9-month follow-ups
Shannon diversity index of oral and gut microbiota at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Oral and gut microbiota will be analyzed from stool, plaque and salivary sample. The diversity of the oral and gut microbiota samples will be measured by the Shannon diversity index.
Concentration of short chain fatty acid in stool samples at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Fecal metabolites will be measured through the concentration of short chain fatty acid in stool samples
3-day food record at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Dietary intake will be assessed using a 3-day food record to determine meal patterns, including macronutrient intake, energy intake, and meal timing
Chinese version of Chrono-nutrition Profile Questionnaire at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Chrono-nutrition behaviors will be evaluated using the Chinese version of the Chrono-nutrition Profile Questionnaire (CP-Q), which includes six distinct aspects: breakfast skipping, timing of the largest meal, evening eating habits, evening latency, nighttime eating behaviors, and eating window.
Chinese version of Munich Chronotype Questionnaire at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Chronotype will be assessed by Chinese version of Munich Chronotype Questionnaire (MCTQ). The computed variables of workdays and work-free days from this questionnaire include sleep onset (SOw, SOf, hh:mm), local time of getting out of bed (GUw, GUf, hh:mm), sleep duration (SDw, SDf, hh:mm), total time in bed (TBTw, TBTf, hh:mm), mid-sleep (MSW, MSF, hh:mm). The computation of the variables include: Average weekly sleep duration (hh:mm) =(SDw x WD + SDf x FD)/7, Chronotype (hh:mm) =If SDf ≤ SDw: MSF; If SDf > SDw: MSF - (SDf - SDweek)/2, Weekly sleep loss (hh:mm) = If SDweek > SDw: (SDweek - SDw) x WD; If SDweek ≤ SDw: (SDweek - SDf) x FD, Relative social jetlag (hh:mm) = MSF - MSW, Absolute social jetlag (hh:mm) = | MSF - MSW |, Average weekly light exposure (hh:mm) = (LEw x WD + LEf x FD)/7
Chinese version of international physical activity questionnaire short form at baseline, 3-month and 9-month follow-ups | at baseline, 3-month and 9-month follow-ups
  Physical activity (PA) levels will be evaluated by a Chinese version of international physical activity questionnaire short form (IPAQ). Total PA (min/wk) = 2x time spent on vigorous + moderate + walking, MET (Metabolic Equivalent of Task, min/wk) = 8 x vigorous +4x moderate + 3.3 x walking

CONTACTS AND LOCATIONS:
Overall Officials: Walter Y.H. Lam, Prof., Principal Investigator — The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, Sai Ying Pun, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided